CLINICAL TRIAL: NCT00166062
Title: Safety and Effectiveness of Computer Screening for Intimate Partner Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Debra Houry, MD, MPH, Principal Investigator, Emory University
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 0304-2003; R49/CCR423113-03 (Other: Other)
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Domestic Violence; Perpetration
Keywords: intimate partner violence; perpetration
MeSH Terms: interventions — Poliovirus Vaccine, Inactivated

INTERVENTIONS:
Procedure: Screening patients for IPV

SUMMARY:
The purpose of this study is to see if using a computer kiosk to screen men and women for intimate partner violence victimization and perpetration is safe and effective. We hypothesize that screening will not result in any adverse events.

DETAILED DESCRIPTION:
All eligible ER patients will be screened during study times for IPV victimization and perpetration. All victims will be followed at 1 week and 3 months to determine any adverse outcomes. Perpetrators will only be followed in the ED for adverse outcomes after screening. All patients who disclose IPV victimization or perpetration will get a list of community resources. Victims will be asked at follow up what resources they used.

ELIGIBILITY:
Inclusion Criteria: Men and women age 18-55 who present to the emergency department waiting room during study hours

-

Exclusion Criteria:

* Acutely intoxicated, psychotic, unable to read, not English speaking

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Dates: Start 2004-01; Primary Completion 2006-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Adverse events in the ED
Increased violence at follow up

CONTACTS AND LOCATIONS:
Overall Officials: Debra Houry, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States